CLINICAL TRIAL: NCT03361124
Title: Oxytocin Dosing at Planned Cesarean Section and Postpartum Anemia: A Comparison of Two Protocols
Brief Title: Oxytocin Dosing at Planned Cesarean Section and Anemia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator no longer interested in proceeding with study
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Helana Pietragallo, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00006502
Record Dates: First submitted 2017-08-01; First posted 2017-12-04 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Blood Loss Anemia; Uterine Atony With Hemorrhage
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded controlled
Who Masked: Participant, Investigator
Masking Description: Covering of labels on IV fluids
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Patient will receive standard post-partum Oxytocin (20 mU in 1 L LR) and 1 L LR over 8 hours following delivery.
  Interventions: Drug: Oxytocin
- Treatment (Experimental): Patient will receive standard post-partum Oxytocin(20 mU in 1 L LR) an additional 20 mU Oxytocin in 1 L LR over 8 hours following delivery.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Administration of additional 20 mU Oxytocin
  Other Names: Pitocin

SUMMARY:
Patient's with planned cesarean sections will be randomized to receive either standard 20 mU in 1L as a bolus following delivery of the placenta or 20 mu in 1L following delivery of the placenta plus an additional 20 mU in 1L over 8 hours.

DETAILED DESCRIPTION:
The purpose of this study is to examine the impact of differential dose protocols commonly utilized in the post cesarean period to determine if laboratory definitions of anemia are different. Oxytocin is an antidiuretic hormone that is utilized after delivery of the fetus and placenta to contract the uterus and decrease blood loss both at the time of surgery and in the post-partum period. Here at the Penn State Hershey Medical center the investigators will use 20 units of oxytocin in a 1 L bag of LR in bolus fashion after delivery of the placenta. Other protocols use an extended course of therapy using 20 units of oxytocin in a 1 L bag of LR in a bolus plus an additional 20 units of oxytocin in a 1 L bag of LR over an 8 hour period of time.

We hypothesize that:

* Women who receive the standard 20 mU of oxytocin in 1L of LR in bolus fashion plus 20 mU in 1L over 8 hours will have a decreased reduction in pre-operative vs post-operative hematocrit and hemoglobin versus those that receive 20 mU in 1L of LR.
* Women who receive the standard 20 mU of oxytocin in 1L of LR in bolus fashion plus 20 mU in 1L over 8 hours will have decreased blood loss by weight in the postpartum period compared to patients who receive 20 mU in 1L of LR.

ELIGIBILITY:
Inclusion Criteria:

* Planned cesarean sections for singletons at or greater than 37 weeks gestational age
* Primary or repeat cesarean section will be included

Exclusion Criteria:

* Multiple fetal pregnancies
* Hematologic disorders
* Fetal anomalies
* Pre-eclampsia. These patients are at increased risk of fluid overload and so fluid status may be affected by receiving a second bag of fluid containing oxytocin in the postpartum period.
* Known contraindication to oxytocin
* Hypersensitivity to oxytocin
* Patients who have labored and then proceed with cesarean section for any reason. Patients who have labored have had either intrinsic or extrinsic exposure to oxytocin. These patients may have decreased sensitivity to oxytocin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Blood loss in postpartum period defined by grams/hour | 3-4 days after delivery
  Measure pads used post-partum

SECONDARY OUTCOMES:
Change in Hemoglobin | 24 hours
  Pre-op hemoglobin and post-op hemoglobin
Change in Hematocrit | 24 hours
  Pre-op hematocrit and post-op hematocrit
Length of hospital stay | 3-4 days after delivery
  Start of surgery to discharge (hours)
Need for additional uterotonics | 24 hours after delivery
  Use of uterotonics
Continuation of breastfeeding | 6 weeks
  Is patient breastfeeding at 6 week post-partum visit
Quantity of narcotic pain medications | 3-4 days after delivery
  Number of narcotic tablets used from time of surgery to discharge
Attendance at post-partum visit | 6 weeks
  Did patient attend post-partum visit?
Post-partum complications | 6 weeks
  Did patient have surgical wound infection, endometritis?
Need for blood transfusion | 3-4 days after delivery
  Did the patient require blood transfusion?
Edinburgh post-partum depression scale >10 | 6 weeks
  Did the patient score greater than 10 points on Edinburgh post-partum depression scale?

CONTACTS AND LOCATIONS:
Overall Officials: Helana Pietragallo, MD, Principal Investigator — Penn State College of Medicine

IPD SHARING:
Plan to Share IPD: Undecided